CLINICAL TRIAL: NCT05014373
Title: An Investigation of the Efficacy and Safety of Favipiravir in Hospitalized NON- SEVERE COVID-19 Patients - An Open-label Randomized Controlled Multi Center Trial
Brief Title: Philippine Trial to Determine Efficacy and Safety of Favipiravir for COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Philippines (Other)
Collaborators: Department of Health, Philippines (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJREB 2020-34
Record Dates: First submitted 2021-06-14; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Favipiravir + Best supportive Care (Active Comparator): Favipiravir (or Avigan) 1800 mg tablet 2x a day on Day 1 then 800 mg 2x a day from Day 2 to maximum of Day 14
  Interventions: Combination Product: Favipiravir + Standard of Care; Procedure: Standard of Care
- Comparator: Best Supportive Care (Placebo Comparator): Best supportive care or Standard Treatment includes oral or intravenous rehydration, electrolyte correction, antipyretics, analgesics, antibiotics and antiemetic drugs & the medication any patient is on due to any concomitant diseases
  Interventions: Combination Product: Favipiravir + Standard of Care; Procedure: Standard of Care

INTERVENTIONS:
Combination Product: Favipiravir + Standard of Care — 1800 mg twice daily for one day, followed by 800mg (4 tablets) twice daily
  Plus Standard of Care
Procedure: Standard of Care — Best supportive care includes Standard treatment included oral or intravenous rehydration, electrolyte correction, antipyretics, analgesics, antibiotics and antiemetic drugs & the medication any patient is on due to any concomitant diseases.

SUMMARY:
This is an open label randomized controlled clinical trial which was designed to confirm the potential efficacy and safety of favipiravir in the management of patients with mild to moderate COVID-19 compared to best supportive care.

DETAILED DESCRIPTION:
Favipiravir is an antiviral agent whose indication in Japan is currently for influenza infections. There were earlier reports from China suggesting its promising potential for benefit in the treatment of COVID-19. This is an open label randomized controlled clinical trial was designed to verify the potential efficacy and safety of favipiravir in the management of patients with mild to moderate COVID-19 compared to best supportive care. This study will look at the potential of using this repurposed oral agent in managing non-severe cases of COVID19. Consenting patients admitted to hospitals or isolation/quarantine facilities will be randomized at a 2:1 ratio to either favipiravir versus best supportive care. Patients will be examined daily and will have xray and nasopharyngeal swabs every 3-4 days for close monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 74 years (at the time of informed consent)
* Gender: Male or female
* Patients with SARS-CoV-2-positive nasopharyngeal swab by RT-PCR test with non-severe presentation upon admission to clinical trial site hospitals or trial-supervised quarantine facilities or under trial -supervised home isolation;
* For premenopausal female patients, patients who have been confirmed to be negative on a pregnancy test before administration of the study drug;
* Patients who understand the contents of this study and can provide written consent by themselves without assistance, or as appropriate with their assent and consent of their parents

Exclusion Criteria:

* Patient has manifestation that meets case definition of Severe COVID-19: Adult with clinical signs of pneumonia (fever, cough, dyspnea, fast breathing) plus one of the following: respiratory rate > 30 breaths/min; severe respiratory distress; or SpO2 < 90% on room air.
* Fever (37.5°C) more than 7 days after the onset of fever
* Patients with suspected concomitant bacterial infections (e.g. 1 ng/ml or higher procalcitonin, etc.) prior to initiation of study drug
* Patients with suspected concomitant fungal infections (e.g. 30 pg/ml or higher (1-3)-β-d-glucan, etc.) prior to initiation of study drug
* Patients with suspected concurrent congestive heart failure (e.g. 100 pg/mL or higher NT-pro BNP levels, etc.) prior to initiation of study drug
* Patients with severe hepatic impairment (>Grade 3: ALT >10 times of upper normal limit)
* Patients with renal impairment requiring dialysis
* Patients with disturbed consciousness such as disturbed orientation
* Pregnant or possibly pregnant patients
* Female patients who are unable to consent to contraceptive use of oral contraceptives, mechanical contraceptives such as intrauterine devices or barrier devices (pessaries, condoms), or a combination of these devices during the 7 days after the start of favipiravir administration.
* Male patients whose partner cannot agree to use the contraception method described in (10) above
* Patients who cannot consent to the use of condoms from the start of favipiravir administration to 7 days after the end of favipiravir administration
* Patients with hereditary xanthinuria
* Patients who have previously ever been diagnosed with hypouricemia (< 1 mg/dL) or xanthine urinary calculi
* Patients with a history of gout or on treatment for gout or hyperuricemia
* Patients receiving immunosuppressants
* Patients who received interferon-alpha or drugs with reported antiviral activity against SARS-CoV-2 (hydroxychloroquine sulfate, chloroquine phosphate, lopinavir-ritonavir combination, ciclesonide, nafamostat mesylate, camostat mesylate) within 9 days after fever (37.5°C or more).
* Patients in whom this episode of infection is a recurrence or reinfection of SARS-CoV-2 infection
* Patients who have previously received favipiravir (T-705a)
* Other patients judged ineligible by the principal investigator or sub-investigator

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Time from initiation of treatment to clinical improvement | 4 to 28 days
  The duration from start of treatment (Favipiravir + Standard of care compared to Standard of care) to clinical improvement and maintained for at least 48 hours.
  Criteria for clinical improvement include all three must be reached:
  Body temperature: axillary ≤37.4°C
  Oxygen saturation measured by pulse oximeter of >96% without oxygen inhalation
  Chest imaging findings with changes showing improvement

SECONDARY OUTCOMES:
Clinical effect of Favipiravir + Standard of Care compared to Standard of Care on patient status as measured by 7-point scale | 4 to 14 days of therapy
  Change in the study specific seven-point scale from initiation of treatment to end of treatment
Number of participants with conversion to negative level of SARS-COV2 viral genome | 4 to 14 days of therapy
  Number of participants with conversion to negative level of SARS-COV2 viral genome
Number of participants with Changes in NEWS (National Early Warning Score) | 4 to 14 days of therapy
  Number of participants with Changes in NEWS (National Early Warning Score)
Number of participants with improvement in chest imaging findings | 4 to 14 days of therapy
  Number of participants with improvement in chest imaging findings

CONTACTS AND LOCATIONS:
Overall Officials: Regina. Berba., MD, Principal Investigator — Philippine General Hospital, Manila Philippines
Locations (1):
- Dr. Regina Berba, Manila, National Capital Region, Philippines